CLINICAL TRIAL: NCT06080113
Title: Cancer of the Prostate Treated With Focal Implantation of a RadioactivE Source - The Introduction of Prostate Cancer Targeted Focal Therapy Treatment in Denmark
Brief Title: Cancer of the Prostate Treated With Focal Implantation of a RadioactivE Source
Acronym: CAPFIRE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Lars Boesen, MD, PhD, DMSci, Associate Professor, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22046020
Record Dates: First submitted 2023-04-24; First posted 2023-10-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: MRI; Biopsy; Brachytherapy; Focal treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Curative targeted focal brachytherapy treatment for localized unifocal prostate-cancer
  Interventions: Radiation: Focal Brachytherapy

INTERVENTIONS:
Radiation: Focal Brachytherapy — Targeted focal brachytherapy is an image-guided technique, where the radioactive source is placed only, and directly into the cancerous area of the prostate. The aim is to preserve the normal surrounding prostate gland tissue to limit treatment-related side effects to the adjacent anatomical structures. A multiparametric prostate MRI is used to identify, localize, and delineate the intraprostatic PCa tumour lesion and plan treatment. A specialized MRI-ultrasound image-fusion software combines the MRI-images with dynamic ultrasound performed in the operating room and is used to focally guide the placement of the radioactive source in the prostate cancer (PCa) tumour focus based on focal dosimetry calculations. A safety margin around the tumour is applied where it is possible to account for MRI tumour volume underestimation, microscopic spread, and treatment uncertainties.

SUMMARY:
The purpose is to assess and describe the oncological and functional outcomes following the introduction of curative targeted focal brachytherapy of prostate cancer in Denmark.

Men with a single MRI-identifiable prostate cancer index-tumour who fulfil inclusion criteria and are candidates for curative treatment. Eligible men will undergo curative intended targeted focal brachytherapy for treatment of histologically confirmed prostate cancer.

The intervention will include Low- (LDR) or High (HDR) dose rate targeted focal brachytherapy of prostate cancer. Collection of data on safety, morbidity, side effects and quality of life. Collection of clinical data on treatment efficacy, progression, and mortality.

All patients will have a follow up of 10-years for oncological outcome, 5-years for acute- and late toxicity-, and 2-years for functional outcomes, respectively. The follow up will include clinical data, MRI, confirmatory biopsies, and questionnaires at specific fixed time points pre-and post-operatively after 1-3 days, 4-weeks, 3-, 6--, 9-, 12-, 18-, and 24-months followed by every 6 months up to 5-yr and then every year up to 10-yr follow-up.

Anticipated number of patients is 50 and regular analysis and reporting will be performed continuously. The first short-term analysis will be after 18-months of follow-up after confirmatory MRI and biopsies, and the final reporting will be after 10-years follow-up in 2035.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80; Performance status 0-1; >10 yr. life expectancy
* Candidate for curative intended treatment
* PSA <20 ng/mL
* Clinical stage T1c or T2a
* Prostate anatomy suitable for focal brachytherapy
* MRI identified index tumour (PI-RADS 3-5) with PCa confirmed on biopsy
* A single index tumour focus with Gleason score 6 (>10 mm maximum cancer-core length [MCCL]), Gleason score 3+4 (any MCCL) or Gleason core 4+3 (<10 mm MCCL)
* Systematic biopsies (≥10-12 cores) with no or low volume Gleason score 6 (3+3) PCa only
* No severe urinary obstructive symptoms (e.g., urinary retention needing indwelling catheter)
* Fit to undergo all procedures in the protocol
* Included subjects should be able to participate in the planned follow-up (either on-site visits or telephone consultation accepted at specific time-points).
* Included subjects should be able to read and understand the study details, and provide written informed consent to participate

Exclusion Criteria:

If any of the following criteria is present, the subject cannot participate in the study:

* Not a candidate for curative intended treatment (e.g., other active malignancy except for non-melanoma skin-cancer, life-expectancy <10 years, severe comorbidities etc.)
* Prior surgical or radiation treatment of PCa; Prior transurethral-resection (TUR-P) is not an exclusion criterion.
* Evidence/suspicion of extra prostatic extension on MRI
* Tumour focus >50% of one prostate half on MRI corresponding to stage >T2a
* Briganti 2018 score ≥7%
* PCa with intraductal carcinoma, cribriform pattern, or small cell component
* Any anatomical or clinical conditional not suitable for brachytherapy (e.g., imperforate anus, prostatitis, inflammatory bowel disease, severe calcifications etc.)
* Any contraindication for prostate MRI (e.g., claustrophobia, pacemaker, estimated glomerular filtration rate ≤30 mL/min/1.73m2)
* Reduction in MRI image quality that interferes with diagnosis caused by e.g., hip replacement surgery or other metal implants in the pelvic area.
* Any medical condition precluding procedures
* Any medication that may alter prostate morphology or alter MRI appearance (e.g., 5-alpha reductase inhibitors, prior androgen deprivation therapy [ADT])
* Subjects who are unwilling or unable to adhere to the study requirements (including treatment, required assessments and follow-up).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with local treatment control at 18-month post treatment | 18 months
  An MRI followed by targeted prostate biopsies are performed 18 months post-treatment.
  Lack of pathological control (progression) is defined by:
  * No pathological changes on biopsy from baseline (stable disease); and/or
  * Tumour upgrading (increase in maximum cancer core length (measured in mm) or higher-grade tumour with increasing Gleason grade (aggressiveness score 1-5, where 5 is worst) compared to baseline.
  These two measurements will be aggregated to arrive at one reported value for the question:
  - Pathological control at 18-month post treatment (yes/no).

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events | 24-months post treatment
  Adverse events are assessed by
  • CTCAEv5 (Common Terminology Criteria for Adverse Events) changes from baseline to post-treatment; Grading 0-5. Higher scores mean worse outcome
  The CTCAEv5 will be assessed before treatment, 1-3 days postoperatively, and at routine post-treatment follow-up visits (see below) up to two years following treatment, or at any time upon withdrawal or pathological or biochemical failure.
Number of patients with treatment related urinary dysfunction | 24-months post treatment
  Adverse events are assessed by
  • IPSS (International Prostate Symptom Score) changes from baseline to post-treatment; Grading 0-35.Higher scores mean worse outcome
  The abovementioned toxicity-questionnaire will be assessed before treatment, 1-3 days postoperatively, and at routine post-treatment follow-up visits (see below) up to two years following treatment, or at any time upon withdrawal or pathological or biochemical failure.
Number of patients with treatment related erectile dysfunction | 24-months post treatment
  Adverse events are assessed by
  • IIEF-5 questionnaire (International Index of Erectile Dysfunction) changes from baseline to post-treatment; Grading 5-25. Higher scores mean worse outcome
  The abovementioned questionnaire will be assessed before treatment, 1-3 days postoperatively, and at routine post-treatment follow-up visits (see below) up to two years following treatment, or at any time upon withdrawal or pathological or biochemical failure.
Number of patients with treatment related bowel dysfunction | 24-months post treatment
  Adverse events are assessed by
  • EPIC bowel domain questionnaire (Extended Prostate Cancer Index - Bowel function) changes from baseline to post-treatment; Grading 0-24.Higher scores mean worse outcome
  The abovementioned questionnaire will be assessed before treatment, 1-3 days postoperatively, and at routine post-treatment follow-up visits (see below) up to two years following treatment, or at any time upon withdrawal or pathological or biochemical failure.
Number of patients with treatment related quality of life changes | 24-months post treatment
  Adverse events are assessed by
  SF-12 v2 questionnaire (Short Form Quality of life assessment) changes from baseline to post-treatment; Grading 12-56.Higher scores mean worse outcome
  The abovementioned questionnaire will be assessed before treatment, 1-3 days postoperatively, and at routine post-treatment follow-up visits (see below) up to two years following treatment, or at any time upon withdrawal or pathological or biochemical failure.
Number of patients with clinical progression at 3-, 5- and 10-yrs | 10 years post-treatment
  Clinical progression can be defined as either biochemical- or pathological progression. Biochemical progression is defined as prostate-specific-antigen (PSA) increase >2 over nadir with an increase >0.75 ng/ml per year. PSA levels will be analyzed prior to routine post-treatment follow-up visits. First appointment is planned at 4 weeks following treatment, then three-monthly for 12 months, six-monthly up to five years post treatment, then yearly until ten years following treatment, or at any time upon withdrawal. In case of biochemical failure, a repeat MRI + biopsies are performed. Due to potential risk of PSA fluctuations ("PSA bounce") during the first 18-24 months following implantation, biochemical progression will not be defined before the primary outcome has been assessed 18 months post-treatment. Secondary definitions of biochemical failure such as PSA-density nadir + 0.1 ng/mL/cc will be analyzed. Pathological progression is defined as under primary outcome.
Rate of salvage treatment | 10 years post-treatment
  The rate of salvage therapy is defined by the percentage of men who receive salvage treatment because of local disease progression following targeted focal brachytherapy. Salvage therapy may include (but not limited to) whole-gland radical prostatectomy, external beam radiation therapy, or re-treatment using focal brachytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Boesen, MD,PhD,DMSci, Principal Investigator — Department of Urology
Locations (1):
- Department of Urology, Herlev University Hospital Herlev, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No